CLINICAL TRIAL: NCT06807879
Title: EFFECTS of OTAGO EXERCISES in ADDITION to ROUTINE PHYSICAL THERAPY on BALANCE and FUNCTIONAL ACTIVITIES in PATIENTS with STROKE.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Affaf Abid, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC-UOL-/380/08/24
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Balance; Ischemic Stroke; Function; OEP
Keywords: Otago Exercise; Functional Activities; Balance; Ischemic Stroke; Physical therapy
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: GROUP A :Modified Otago Exercise with Routine care Physical therapy GROUP B :Routine Care Physical Therapy
Who Masked: Outcomes Assessor
Masking Description: Single-blinded assessor was considered to minimize bias in outcome measurements. The assessor was unaware of the intervention group assignment for each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified Otago Exercise with Routine care Physical therapy (Experimental): The modified-OEP group intervention consisted of 15 min of walking followed by a 30 min Otago Exercise Program consisting of balance and strength training, followed by another 15 min of walking. The 15 min walking was accomplished through continuous walking at an individual pace in the ~15 m training room. Participants were asked to walk 15 m, make a U-turn towards the left side, walk 15 m, then make a U-turn towards the right side at the next turning point, in order to achieve an equivalent effect on the promoted benefit of symmetry when turning left and right. This was repeated until the session was complete.
  Interventions: Behavioral: Modified Otago Exercise with Routine care Physical therapy
- Routine Care Physical Therapy (Experimental): The routine care physical therapy session typically involves a variety of exercises aimed at general strengthening, stretching, and basic gait training. 1 hour of standard physiotherapy exercises focusing on general strengthening, stretching, and basic gait training.
  Interventions: Behavioral: Routine Care Physical Therapy

INTERVENTIONS:
Behavioral: Modified Otago Exercise with Routine care Physical therapy — To improve the efficacy of the balance improvement intervention, we modified the OEP by incorporating the additional walking, recommended by the OEP guidelines, into a single exercise session and conducting it as a group exercise program in accordance with a previous meta-analysis (Chiu et al., 2021) . As shown in Figure 1, the modified-OEP group intervention consisted of 15 min of walking followed by a 30 min Otago Exercise Program consisting of balance and strength training, followed by another 15 min of walking. The 15 min walking was accomplished through continuous walking at an individual pace in the ~15m training room. Participants were asked to walk 15 m, make a U-turn towards the left side, walk 15 m, then make a U-turn towards the right side at the next turning point, in order to achieve an equivalent effect on the promoted benefit of symmetry when turning left and right.
  This was repeated until the session was complete.
  Arms: Modified Otago Exercise with Routine care Physical therapy
Behavioral: Routine Care Physical Therapy — The routine care physical therapy session typically involves a variety of exercises aimed at general strengthening, stretching, and basic gait training. 1 hour of standard physiotherapy exercises focusing on general strengthening, stretching, and basic gait training. The session included a combination of exercises aimed at general strengthening, such as core stability exercises, muscle-strengthening exercises with weights or resistance bands and functional movements like squats and lunges. Stretching exercises targeting key muscle groups like hamstrings will be incorporated to improve flexibility and range of motion. Gait training will focus on activities like side lunges, step-ups, and balance exercises to enhance walking ability and postural control. Additionally, the plan emphasized progressive challenges incorporating a mix of static and dynamic balance exercises using tools like foam pads or balance boards.
  Arms: Routine Care Physical Therapy

SUMMARY:
Stroke is an extremely severe medical condition which is ranked as the second biggest cause of death worldwide as it claims an estimated 5.5 million lives per year. A stroke can result in enduring brain injury, prolonged disability, or fatality (Tsao et al., 2023) . There are two major types of stroke: Hemorrhagic stroke and Ischemic stroke. The most prevalent type is Ischemic, accounting for approximately 87% of strokes worldwide. It arises from a blockage in a blood vessel supplying the brain (Collaborators, 2022) . Also, the affected brain areas can result in functional limitations, cognitive changes, and emotional difficulties (Fihla, 2024) .

Moreover, given the potential cost-effectiveness of OEP compared to more intensive rehabilitation methods, its implementation could offer a pragmatic solution to improving the quality of life for individuals grappling with the enduring consequences of ischemic stroke.

Therefore, exploring the effectiveness of OEP in this specific population holds promise for advancing stroke rehabilitation strategies and potentially improving the lives of individuals living with the long-term effects of ischemic stroke.

DETAILED DESCRIPTION:
Study Design: Randomized Clinical Trial.

Screening:

Patients were screened to meet inclusion criteria. The consent form taken from patients then patients were randomly allocated into two groups ( 29 in each group).

Randomization:

Using the lottery approach, patients who met the inclusion criteria were split into experimental and control groups at random by the online tool for randomization.

Blinding:

To ensure precision and mitigating the bias the assessor of outcome was kept blind also. An independent assessor specialized in this technique and having more than 5 years experience screened patients, and they were subsequently randomly assigned to either the experimental group. The computer-generated allocation sequence was established prior to the study's commencement.

Assessment:

Data was collected at baseline, fourth week and then at the end of the eighth week. Baseline assessments will be conducted before the intervention. Post-intervention assessments will be conducted immediately after the intervention. Statistical analysis will include descriptive statistics, t-tests, and analysis of variance to compare the outcomes between the two groups.

Intervention:

The intervention group A received routine physical therapy in addition to the Otago Exercise Program, while the control group B received routine physical therapy alone.

GROUP A: ( Modified Otago Exercise with Routine care Physical therapy) GROUP B: ( ROUTINE CARE PHYSICAL THERAPY )

Outcome Measures:

Primary outcome:

Balance was assessed using the Berg Balance Scale (BBS)

Secondary outcomes:

Functional activities the physical performance was assessed using the 30-s Chair Stand Test (30 s-CST).

Ethical Considerations: This study has received ethical approval from the Institutional Review Board (IRB). Informed consent was obtained from all participants.

Data Analysis: Statistical software was used to analyze the data, with appropriate tests employed based on data normality to compare outcomes between groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 60 to 70 years old (Verheyden et al., 2013).
* Both genders (Khumpaneid et al., 2022).
* Patients who have been diagnosed with ischemic stroke by a medical professional(Khumpaneid et al., 2022).
* Eligible for movement without using any walking aid equipment (Khumpaneid et al.,2022).
* Exercise less than 150 mins per week (Khumpaneid et al., 2022).
* Timed Up and Go score is more than 10 (Khumpaneid et al., 2022).
* Mini-Mental State Examination (MMSE) score ≥ 24 (Page et al., 2007).
* Urinary and bowel continence (Jin et al., 2023) .

Exclusion Criteria:

* Patients who have severe cognitive impairment or communication difficulties (Jin et al., 2023).
* Participants who have neurological conditions (e.g., Parkinson's disease), vision problems or contagious diseases (Khumpaneid et al., 2022).
* Patients who have undergone surgery in the past 3 months (Jin et al., 2023

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Balance | Baseline, mid-intervention (4 weeks), and post-intervention (8 weeks).
  Balance was assessed using the Berg Balance Scale (BBS). To determine the effects of Otago exercises in addition to routine physical therapy on balance and functional activities in patients with stroke.

SECONDARY OUTCOMES:
Functional activities | Baseline, mid-intervention (4 weeks), and post-intervention (8 weeks).
  Functional activities was assessed using the 30-s Chair Stand Test (30 s-CST).

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Saghir, MS Neuro, Principal Investigator — University of Lahore; Sana Ikram, MS MSK, Study Director — University of Lahore
Locations (1):
- University Of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khumpaneid N, Phoka T, Khongprasert S. Effects of Modified-Otago Exercise Program on Four Components of Actual Balance and Perceived Balance in Healthy Older Adults. Geriatrics (Basel). 2022 Aug 30;7(5):88. doi: 10.3390/geriatrics7050088. PMID 36136797
- [Background] Hatem SM, Saussez G, Della Faille M, Prist V, Zhang X, Dispa D, Bleyenheuft Y. Rehabilitation of Motor Function after Stroke: A Multiple Systematic Review Focused on Techniques to Stimulate Upper Extremity Recovery. Front Hum Neurosci. 2016 Sep 13;10:442. doi: 10.3389/fnhum.2016.00442. eCollection 2016. PMID 27679565
- [Background] Farooq A, Venketasubramanian N, Wasay M. Stroke Care in Pakistan. Cerebrovasc Dis Extra. 2021;11(3):118-121. doi: 10.1159/000519554. Epub 2021 Oct 25. PMID 34695824
- [Background] Everard G, Luc A, Doumas I, Ajana K, Stoquart G, Edwards MG, Lejeune T. Self-Rehabilitation for Post-Stroke Motor Function and Activity-A Systematic Review and Meta-Analysis. Neurorehabil Neural Repair. 2021 Dec;35(12):1043-1058. doi: 10.1177/15459683211048773. Epub 2021 Oct 25. PMID 34696645
- [Background] Davis JC, Khan KM, Hsu CL, Chan P, Cook WL, Dian L, Liu-Ambrose T. Action Seniors! Cost-Effectiveness Analysis of a Secondary Falls Prevention Strategy Among Community-Dwelling Older Fallers. J Am Geriatr Soc. 2020 Sep;68(9):1988-1997. doi: 10.1111/jgs.16476. Epub 2020 May 29. PMID 32472567
- [Background] Davis JC, Hsu CL, Barha C, Jehu DA, Chan P, Ghag C, Jacova P, Adjetey C, Dian L, Parmar N, Madden K, Liu-Ambrose T. Comparing the cost-effectiveness of the Otago Exercise Programme among older women and men: A secondary analysis of a randomized controlled trial. PLoS One. 2022 Apr 20;17(4):e0267247. doi: 10.1371/journal.pone.0267247. eCollection 2022. PMID 35442974
- [Background] Angeles CM, Laura AM, Consuelo CM, Manuel RR, Eva AC, Covadonga GA; Otago Project Working Group. The effect that the Otago Exercise Programme had on fear of falling in community dwellers aged 65-80 and associated factors. Arch Gerontol Geriatr. 2022 Mar-Apr;99:104620. doi: 10.1016/j.archger.2022.104620. Epub 2022 Jan 4. PMID 34999543
- [Background] Ambrosini E, Peri E, Nava C, Longoni L, Monticone M, Pedrocchi A, Ferriero G, Ferrante S. A multimodal training with visual biofeedback in subacute stroke survivors: a randomized controlled trial. Eur J Phys Rehabil Med. 2020 Feb;56(1):24-33. doi: 10.23736/S1973-9087.19.05847-7. Epub 2019 Sep 26. PMID 31556542
- [Background] Alsubiheen AM, Choi W, Yu W, Lee H. The Effect of Task-Oriented Activities Training on Upper-Limb Function, Daily Activities, and Quality of Life in Chronic Stroke Patients: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Oct 29;19(21):14125. doi: 10.3390/ijerph192114125. PMID 36361001
- [Background] Albornos-Munoz L, Moreno-Casbas MT, Sanchez-Pablo C, Bays-Moneo A, Fernandez-Dominguez JC, Rich-Ruiz M, Gea-Sanchez M; Otago Project Working Group. Efficacy of the Otago Exercise Programme to reduce falls in community-dwelling adults aged 65-80 years old when delivered as group or individual training. J Adv Nurs. 2018 Jul;74(7):1700-1711. doi: 10.1111/jan.13583. Epub 2018 Jun 3. PMID 29633328
- [Background] Ahmed, S., Manzoor, F., Naseem, H., & Ansari, A. Q. (2024). Effects of action observation therapy with Otago exercises on balance and quality of life in older adults. The Rehabilitation Journal, 15-21.